CLINICAL TRIAL: NCT02480387
Title: A Phase 2, Single-Center, Open-Label Pilot Study to Investigate the Efficacy and Safety of Sofosbuvir/Ledipasvir Fixed-Dose Combination for 8 Weeks in Subjects With Chronic Genotype 1 Hepatitis C Virus (HCV) and Human Immunodeficiency Virus (HIV)-1 Coinfection
Brief Title: Efficacy and Safety of Ledipasvir/Sofosbuvir Fixed-Dose Combination for 8 Weeks in Subjects With Chronic Genotype 1 HCV and HIV-1 Co-infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peter J. Ruane, M.D., Inc. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IN-US-337-1821
Record Dates: First submitted 2015-06-19; First posted 2015-06-24 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-02

CONDITIONS: Treatment of Hepatitis C
MeSH Terms: interventions — ledipasvir; ledipasvir, sofosbuvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment Arm (Experimental): 8 weeks treatment with Ledipasvir/Sofosbuvir FDC
  Interventions: Drug: Ledipasvir/Sofosbuvir FDC

INTERVENTIONS:
Drug: Ledipasvir/Sofosbuvir FDC
  Other Names: Harvoni

SUMMARY:
Target Population: Hepatitis C Treatment Naïve, non-cirrhotic, Chronic genotype 1 hepatitis C virus (HCV) infected adults that are co-infected with human immunodeficiency virus (HIV)-1and have HCV RNA < 6 x106 IU/mL

Duration of Subjects will be treated for 8 weeks and followed for 24 weeks post- Treatment: treatment

ELIGIBILITY:
Inclusion Criteria:

* Chronic HCV GT1, treatment-naïve, non-cirrhotic adult subjects.
* HCV RNA levels more than 10,000 IU/mL and less than 6,000,000 IU/mL at Screening

Exclusion Criteria:

* Gastrointestinal disorder or post-operative condition that could interfere with the absorption of the study drug.
* Solid organ transplantation.
* Significant cardiac disease or other significant co-morbidities that could interfere with study treatment.
* Malignancy within the 3 years prior to screening, with the exception of specific cancers that have been cured by surgical resection (basal cell skin cancer, etc.). Subjects under evaluation for possible malignancy are not eligible.
* Infection with hepatitis B virus (HBV)

Min Age: 18 Years | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-05; Primary Completion 2015-11 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
SVR12 | Sustained Virologic Response 12 Weeks Post-Treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Peter J. Ruane, MD, Inc., Los Angeles, California, United States